CLINICAL TRIAL: NCT01992497
Title: Effect,Tolerance and Safety of a Supplementation With a Probiotic in Healthy Newborn Term Infants Born by Cesarean Section Over a 12 Months Period Study
Brief Title: Cesarean Section Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 12.14.INF
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Diarrhea; Atopic Dermatitis
Keywords: Cesarean section, probiotic, formula fed, gut microbiota
MeSH Terms: conditions — Diarrhea; Dermatitis, Atopic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Formula + placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Probiotic
- Formula + probiotic (Experimental): Formula + probiotic
  Interventions: Dietary Supplement: Probiotic
- Breastfed + probiotic (Experimental): Breastfed + probiotic
  Interventions: Dietary Supplement: Probiotic
- Breastfed + placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic

SUMMARY:
Effect, tolerance and safety of a supplementation with a probiotic on the risk of gastrointestinal infections, on growth, and on gut microbiota in healthy newborn term infants born by Cesarean section. Exploratory comparison between a probiotic vs. placebo in the formula-fed and in the breastfed feeding groups.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent must be obtained from legal guardian(s) prior to randomization or any study related procedures
* healthy newborns
* born by Cesarean section
* singleton birth
* Age at enrollment in the study < 24h
* birth weight ≥ 2500g and ≤ 4300g
* gestational age ≥ 37 weeks and ≤ 42 weeks

Exclusion Criteria:

* congenital diseases or malformations that may inhibit growth
* prenatal and/or postnatal diseases
* parents are expected to have difficulty complying with the feeding regime
* planned re-admittance to the hospital in the first 14 days of life
* antibiotic treatment at the time of enrollment in the study

Ages: 1 Minute to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 721 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of diarrhea episodes between a probiotic vs. placebo | 12 months

SECONDARY OUTCOMES:
Diarrhea duration between a probiotic vs. placebo | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Ernst v. Bergmann GmbH, Potsdam, Germany